CLINICAL TRIAL: NCT06866431
Title: Effect Of Cavitation In Post-Extractive Socket Healing
Acronym: Piezoclean
Status: Recruiting | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, Adjunct Professor, University of Trieste
Other Study IDs: PIEZOCLEAN
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cavitation; Healing of Extraction Socket

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Piezoclean: Ultrasonic cavitation treatment with 0.9% sodium chloride via a specific insert (Piezoclean, Esacrom, Imola, Italy) driven by a piezoelectric device in post extractive socket
  Interventions: Procedure: Piezoclean
- Control: Simple 0.9% sodium chloride irrigation in post extractive socket
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Piezoclean — Following local anesthesia and periotomy, flapless extraction will be performed using forceps and elevators. After socket debridement with Lucas surgical curette, the extraction sockets will be randomly divided into test and control group.Test group sites will receive 90 seconds of ultrasonic cavitation treatment with 0.9% sodium chloride via a specific insert (Piezoclean, Esacrom, Imola, Italy) driven by a piezoelectric device with the following modalities: i) piezo settings: SURGERY 1 U 040 V 080 P 100; ii) no pressure should be applied to prevent the steel insert from coming into contact with the bone; iii) do not create a complete seal to avoid heating the liquid, which could cause potential discomfort or harm to the patient.
  An "X" suture will be then applied using non-resorbable synthetic monofilament.
  Groups: Piezoclean
Procedure: Control — Following local anesthesia and periotomy, flapless extraction will be performed using forceps and elevators. After socket debridement with Lucas surgical curette, the extraction sockets will be randomly divided into test and control group. In control group, a simple 0.9% sodium chloride irrigation (control group) will be performed.
  An "X" suture will be then applied using non-resorbable synthetic monofilament.
  Groups: Control

SUMMARY:
In everyday clinical practice, the proper management of the post-extraction socket is crucial in order to enable an optimal healing of the wound and a close post-surgical monitoring is critical to prevent possible complications. After an injury, the cellular reaction starts early, presenting significant changes as soon as 12 to 24 hours later. Favourable wound healing begins with the timely formation, organization, stabilization, and attachment of the blood clot. The stability of the clot is influenced by various factors including the host response, local anatomical characteristics, presence of bacteria and severity of surgical trauma. Delayed healing can lead to increased complications, patient discomfort, and potential procedure failures. In the light of these considerations, the proven effectiveness of piezoelectric devices to facilitate healing mechanisms is known in literature. Inverse piezoelectric effect, as used in current devices, creates mechanical shock waves that oscillate linearly at sonic and ultrasonic frequencies (from 30 to 30.000 Hz). In addition, mechanical micro-movements with a frequency between approximately 24 and 30 kHz create a cavitation effect in the irrigation solution, limiting intraoperative bleeding, thereby increasing the visibility and safety of the procedure.

The purpose of the present study is to evaluate if the application of cavitation effect of post-extractive socket is capable of reducing healing time and Numeric Pain Rating Scale (NPRS) values.

DETAILED DESCRIPTION:
Methods: Subjects referring to the clinical centers with the clinical indication of extraction of two contralateral single-rooted teeth of the same arch are suitable for enrollment. Teeth to be extracted should be characterized by the following condition: deep unrecoverable decay; untreatable endodontic issue; untreatable crow-root fracture.

The same surgical extractive protocol will be performed in both sites. Following local anesthesia and periotomy, flapless extraction will be performed using forceps and elevators. After socket debridement with Lucas surgical curette, the extraction sockets will be randomly divided into test and control group. Test group sites will receive 90 seconds of ultrasonic cavitation treatment with 0.9% sodium chloride via a specific insert (Piezoclean, Esacrom, Imola, Italy) driven by a piezoelectric device with the following modalities: i) piezo settings: SURGERY 1 U 040 V 080 P 100; ii) no pressure should be applied to prevent the steel insert from coming into contact with the bone; iii) do not create a complete seal to avoid heating the liquid, which could cause potential discomfort or harm to the patient.

In control group, a simple 0.9% sodium chloride irrigation (control group) will be performed.

An "X" suture will be then applied using non-resorbable synthetic monofilament. All patients will be instructed in post-extractive domiciliary care. Paracetamol 1g every 8 hours in case of pain will be prescribed.

Patients will be given a questionnaire to fill out daily, entering a score on the NPRS (from 1 to 10) for 7 days, where a score of 0 indicates "no pain" and a score of 10 indicates "very severe pain", along with the number of paracetamol intakes per day. Follow-ups will be scheduled for day-3, day-7 for suture removal, day-14, day 21 for final check.

On day 3, day 7, day 14 and day 21 the maturation and quality of tissues will be evaluated using a modified version of the Healing Index (HI) that involves 3 scoring levels for each of the 4 parameters considered:

* tissue color (1 = 100% of gingiva pink; 2 ≤ 50% of gingiva red, hyperemic, movable; 3 ≥ 50% of gingiva red, hyperemic, movable);
* color and consistency of the healing tissue (1 = close grained, pink; 2 = soft, red; 3 = fragile, greenish or grayish);
* suppuration (1 = absent; 2 = absent but pronounced amount of plaque around socket walls; 3 = pronounced);
* bleeding (1 = absent; 2 = induced by palpation; 3 = spontaneous). The total score ranged from 4 (excellent healing) to 12 (severely impaired healing).

Study design: Prospective randomized clinical trial.

Study population: The study will be conducted in an outpatient hospital setting.

Subject numerosity: The outcome of the study involves the evaluation of the application of cavitation effect via piezoelectric device on post-extractive sockets.

To date, there are no studies in the literature reporting results regarding the application of cavitation that may be used for an adequate sample size calculation.

Therefore, a minimal clinically important difference (MCID) was considered to be a difference between the means of the group 1 and the group 2 of 0.5 points on NPRS at T1 (3gg), with a standard deviation of 1 point. With alpha set at 0.05 and power set at 0.8, a sample size of 62 statistical units per group was calculated.

Each center will treat 12 patients with bilateral extractions (7 centers = 84 patients), to compensate possible drop-outs during the study.

Enrollment procedure: all patients who meet the inclusion and exclusion criteria will be enrolled in the study following the administration of the Information Sheet and the acquisition of informed consent.

Data collection: Data will be entered in an Excel database, which can be accessed using specific usernames and passwords in the possession of the staff involved in the study. The data will be entered anonymously by associating a numeric ID to each patient.

Data analysis: Statistical analysis will be performed by means of a computerized statistical package (SigmaStat 3.5, SPSS Inc., Germany). Data will be expressed as mean ± SD and median (interquartile range), respectively, for parametric and nonparametric values. Data will be normalized and difference in NPRS between the treatments at the various timepoints will be analyzed with descriptive statistics to assess whether they have a normal distribution; both equal variance and normality tests will be used. Hypotheses will be tested using unpaired t-test in case of normally distributed data, while Mann-Whitney U-test will be performed to compare nonparametric values.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 100 years
* Two single rooted hopeless teeth of the same arch to be extracted
* ASA scale value equal or less than 3
* Signed informed consent

Exclusion Criteria:

* General contraindications for dental and/or surgical treatments
* Inflammatory and autoimmune disease of the oral cavity
* Uncontrolled diabetes (HbA1c > 7.5%)
* History of malignancy requiring chemotherapy or radiotherapy within the past five years
* Previous immunosuppressant bisphosphonate or high dose corticosteroid therapy
* Heavy smokers (> 20 cigarettes /day)
* Pregnancy or lactating women
* No compliance
* Extraction performed after raising a flap and/or with osteotomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with two single rooted hopeless teeth of the same arch to be extracted
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maturation and quality of tissues in post extractive socket | 3 days after tooth extraction
  The maturation and quality of tissues will be evaluated using a modified version of the Healing Index (HI) that involves 3 scoring levels for each of the 4 parameters considered:
  * tissue color (1 = 100% of gingiva pink; 2 ≤ 50% of gingiva red, hyperemic, movable; 3 ≥ 50% of gingiva red, hyperemic, movable);
  * color and consistency of the healing tissue (1 = close grained, pink; 2 = soft, red; 3 = fragile, greenish or grayish);
  * suppuration (1 = absent; 2 = absent but pronounced amount of plaque around socket walls; 3 = pronounced);
  * bleeding (1 = absent; 2 = induced by palpation; 3 = spontaneous). The total score ranged from 4 (excellent healing) to 12 (severely impaired healing).
Maturation and quality of tissues in post extractive socket | 7 days after tooth extraction
  The maturation and quality of tissues will be evaluated using a modified version of the Healing Index (HI) that involves 3 scoring levels for each of the 4 parameters considered:
  * tissue color (1 = 100% of gingiva pink; 2 ≤ 50% of gingiva red, hyperemic, movable; 3 ≥ 50% of gingiva red, hyperemic, movable);
  * color and consistency of the healing tissue (1 = close grained, pink; 2 = soft, red; 3 = fragile, greenish or grayish);
  * suppuration (1 = absent; 2 = absent but pronounced amount of plaque around socket walls; 3 = pronounced);
  * bleeding (1 = absent; 2 = induced by palpation; 3 = spontaneous). The total score ranged from 4 (excellent healing) to 12 (severely impaired healing).
Maturation and quality of tissues in post extractive socket | 14 days after tooth extraction
  The maturation and quality of tissues will be evaluated using a modified version of the Healing Index (HI) that involves 3 scoring levels for each of the 4 parameters considered:
  * tissue color (1 = 100% of gingiva pink; 2 ≤ 50% of gingiva red, hyperemic, movable; 3 ≥ 50% of gingiva red, hyperemic, movable);
  * color and consistency of the healing tissue (1 = close grained, pink; 2 = soft, red; 3 = fragile, greenish or grayish);
  * suppuration (1 = absent; 2 = absent but pronounced amount of plaque around socket walls; 3 = pronounced);
  * bleeding (1 = absent; 2 = induced by palpation; 3 = spontaneous). The total score ranged from 4 (excellent healing) to 12 (severely impaired healing).
Maturation and quality of tissues in post extractive socket | 21 days after tooth extraction
  The maturation and quality of tissues will be evaluated using a modified version of the Healing Index (HI) that involves 3 scoring levels for each of the 4 parameters considered:
  * tissue color (1 = 100% of gingiva pink; 2 ≤ 50% of gingiva red, hyperemic, movable; 3 ≥ 50% of gingiva red, hyperemic, movable);
  * color and consistency of the healing tissue (1 = close grained, pink; 2 = soft, red; 3 = fragile, greenish or grayish);
  * suppuration (1 = absent; 2 = absent but pronounced amount of plaque around socket walls; 3 = pronounced);
  * bleeding (1 = absent; 2 = induced by palpation; 3 = spontaneous). The total score ranged from 4 (excellent healing) to 12 (severely impaired healing).

SECONDARY OUTCOMES:
NPRS | on the day of extraction
  The Numeric Pain Rating Scale (NPRS) is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable.
NPRS | on the first day after extraction
  The Numeric Pain Rating Scale (NPRS) is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable.
NPRS | on the second day after extraction
  The Numeric Pain Rating Scale (NPRS) is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable.
NPRS | on the third day after extraction
  The Numeric Pain Rating Scale (NPRS) is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable.
NPRS | on the fourth day after extraction
  The Numeric Pain Rating Scale (NPRS) is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable.
NPRS | on the fifth day after extraction
  The Numeric Pain Rating Scale (NPRS) is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable.
NPRS | on the sixth day after extraction
  The Numeric Pain Rating Scale (NPRS) is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Trieste, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: No